CLINICAL TRIAL: NCT01225835
Title: Effect of Highly Purified Menotrophin and Recombinant Follicle Stimulating (rFSH, Follitrophin Alpha) in Subfertile Female Patients Undergoing IVF on Progesterone Serum Levels During the Follicular Phase and Their Possible Use as Predictors for the Success Rate of Ongoing Pregnancies
Brief Title: Progesterone Serum Levels in Subfertile Female Patients Undergoing in Vitro Fertilisation (IVF)
Acronym: PREDICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE999906 CS11; 2010-019411-37 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-21 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; Glycoprotein Hormones, alpha Subunit; follitropin alfa; cetrorelix; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; asialogalactochoriongonadotropin; Chorionic Gonadotropin; Progesterone; Crinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menotrophin (Experimental): Starting on Day 2 or 3 of the menstrual cycle, 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
  Interventions: Drug: Menotrophin; Drug: Cetrorelix; Drug: Choriongonadotropin; Drug: Progesterone
- Follitrophin Alpha (Active Comparator): Starting on Day 2 or 3 of the menstrual cycle, 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
  Interventions: Drug: Follitrophin alpha; Drug: Cetrorelix; Drug: Choriongonadotropin; Drug: Progesterone

INTERVENTIONS:
Drug: Menotrophin — Starting on Day 2 or 3 of the menstrual cycle, 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met.
  Other Names: Menogon® HP
  Arms: Menotrophin
Drug: Follitrophin alpha — Starting on Day 2 or 3 of the menstrual cycle, 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met.
  Other Names: Gonal-f®
  Arms: Follitrophin Alpha
Drug: Cetrorelix — Participants self-inject subcutaneously Cetrorelix in the morning at a daily dose of 0.25 mg/day from Day 5 of gonadotrophin administration on and continue throughout the period of gonadotrophin treatment up to day 12 as a maximum. The last dose of Cetrorelix is given on the day of ovulation induction.
  Other Names: Cetrotide®; GnRH antagonist
Drug: Choriongonadotropin — 10,000 IU administered by the Investigator or designated personnel in the evening of the day on which the hCG criterion is met (no later than Day 13). The criterion for hCG administration is three follicles >+17 mm diameter as shown by pelvic ultrasound examination.
  Other Names: Brevactid®; human chorionic gonadotropin (hCG)
Drug: Progesterone — Vaginal gel progesterone is used once daily at a dose of 90 mg for a period of 30 days starting on the day of oocyte retrieval (approximately Day 14).
  Other Names: Crinone®; intravaginal progesterone

SUMMARY:
This study is aimed to demonstrate that highly purified Menotrophin produces significant lower progesterone serum levels during the follicular phase in comparison to Follitropin alpha in the treatment of subfertile females undergoing an in vitro fertilisation (IVF) and to investigate if the progesterone serum levels might be a useful predictor for the success rate of the ongoing pregnancy rates

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subfertile premenopausal female patients eligible for in vitro fertilisation (IVF) treatment
* Aged ≥34 and ≤42 years
* Body mass index of >18 and <28 kg/m^2
* Normal pelvic ultrasound at Screening
* No more than two previous gonadotrophin stimulated cycles of IVF or intracytoplasmic sperm injection (ICSI) in the history of infertility treatment (gonadotrophin stimulated cycles not used for IVF or ICSI do not count; Clomifen cycles are no exclusion criterion)
* At least 3 consecutive ovulatory menstrual cycles of 24-35 days
* No fertility stimulating drugs at all
* Sperm of partner classified as normal according to World Health Organisation (WHO) 2010 criteria
* Clinically normal baseline haematology, clinical chemistry, and urinalysis values
* Negative serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) antibody tests within the last 6 months prior to Screening
* Endocrine test results within the clinically normal limits at Screening

Exclusion Criteria:

* Presence of any clinically relevant systemic disease (e.g., insulin-dependent diabetes mellitus)
* A history of or current endocrine disease (excluding treated hypothyreosis), including polycystic ovary syndrome (PCOS) and hyperprolactinaemia
* A history of coagulation disorders
* Persistent ovarian cysts (>3 months)
* A history of hypersensitivity to any of the constituents of the study medication or related compounds
* Diagnosed poor (<3 oocytes) responders to prior gonadotrophin stimulated ART-cycle
* History of severe ovarian hyperstimulation syndrome in former gonadotrophin stimulated assisted reproductive technology (ART)-cycle

Ages: 34 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (8):
- Germany (8):
  - Fertility Center Berlin, Berlin
  - Praxisklinik Sydow am Gendarmenmarkt, Berlin
  - Kinderwunschzentrum Dortmund, Dortmund
  - Universitätsklinikum Duesseldorf, Frauenklinik, Düsseldorf
  - Praxis für Kinderwunschbehandlung, Erlangen
  - NOVUM Zentrum, Essen
  - IVF Zentrum, Saar
  - Endokrinologikum Ulm, Ulm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred seventy patients were screened.
Groups:
- Menotrophin: Menotrophin 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
- Follitrophin Alpha: Follitrophin alpha 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 12 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
Period: Overall Study
Arm/Group | Menotrophin | Follitrophin Alpha
Started | 62 | 62
Per Protocol Population | 48 | 58
Completed | 55 (hCG criterion met) | 59 (hCG criterion met)
Not Completed | 7 | 3
Not completed — Completed protocol | 2 | 1
Not completed — Did not meet hCG criterion | 2 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Menotrophin | Follitrophin Alpha | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (2.4) | 36.7 (2.3) | 36.6 (2.4)
Age, Customized [Number; unit: participants]
  < 39 years | 50 | 49 | 99
  >=39 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 64.3 (8.2) | 63.5 (8.7) | 63.9 (8.4)
Duration of Infertility [Mean (Standard Deviation); unit: months] | 45.7 (35.0) | 40.6 (25.6) | 43.2 (30.7)
Menstrual Cycle [Number; unit: participants]
  Regular | 62 | 62 | 124
  Irregular | 0 | 0 | 0
Length of Menstrual Cycle [Mean (Standard Deviation); unit: days] | 28.3 (1.7) | 28.2 (1.5) | 28.2 (1.6)
Former Treatment for Infertility [Number; unit: participants]
  No | 24 | 24 | 48
  Yes | 38 | 38 | 76
Participants with Gonadotrophin Stimulated Assisted Reproductive Technology (ART) Cycle [Number; unit: participants]
  No | 0 | 0 | 0
  Yes | 13 | 18 | 31
  Missing Values | 49 | 44 | 93
Aetiology of Infertility [Number; unit: participants]
  Tubal factor | 20 | 18 | 38
  Endometriosis | 4 | 3 | 7
  Idiopathic | 36 | 33 | 69
  Other | 1 | 8 | 9
  Missing values | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Serum Progesterone (P4) Level in the Morning of the Day of Human Chorionic Gonadotrophin (hCG) Administration
Description: Ovulation induction was performed by administration of hCG once three follicles >=17 mm diameter as shown by pelvic ultrasound examination. This outcome compares the serum progesterone level the morning prior to hCG administration across treatment arm, and also by age stratum (<39 years and >=39 years).
Time Frame: approximately day 10
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Menotrophin: Stratum Age <39 Yrs: The subset of participants in the menotrophin treatment arm who were < 39 years old.
- Menotrophin: Stratum Age >=39 Yrs: The subset of participants in the menotrophin treatment arm who were >= 39 years old.
- Follitrophin Alpha: Stratum Age <39 Yrs: The subset of participants in the follitrophin alpha treatment arm who were < 39 years old.
- Follitrophin Alpha: Stratum Age >=39 Yrs: The subset of participants in the follitrophin alpha treatment arm who were >= 39 years old.
Arm/Group | Menotrophin | Menotrophin: Stratum Age <39 Yrs | Menotrophin: Stratum Age >=39 Yrs | Follitrophin Alpha | Follitrophin Alpha: Stratum Age <39 Yrs | Follitrophin Alpha: Stratum Age >=39 Yrs
Number analyzed (Participants) | 62 | 50 | 12 | 62 | 49 | 13
ng/ml | 0.69 (0.34) | 0.72 (0.35) | 0.54 (0.25) | 0.89 (0.41) | 0.92 (0.43) | 0.80 (0.28)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — The significance level is 0.05
Statistical Analysis 2: Comparison: Menotrophin: Stratum Age <39 Yrs vs Follitrophin Alpha: Stratum Age <39 Yrs; Age < 39 years; Test type: Superiority or Other; p = 0.015, t-test, 2 sided — The significance level is 0.05
Statistical Analysis 3: Comparison: Menotrophin: Stratum Age >=39 Yrs vs Follitrophin Alpha: Stratum Age >=39 Yrs; Age >= 39 years; Test type: Superiority or Other; p = 0.027, t-test, 2 sided — The significance level is 0.05

2. Secondary Outcome: Receiver Operating Characteristic (ROC) Analysis of Progesterone as Predictor for Ongoing Pregnancy Rate at Day 7 and Day of hCG Administration
Description: The influence of the progesterone level on the ongoing pregnancy rate (in relation to all randomized patients) was determined by means of the receiver operating characteristic (ROC) curve. Youden's Index (sensitivity + specificity -1) has a range of 0-1, with 0.5 indicating a random effect.
Time Frame: Day 7, approximately Day 10 (hCG Administration)
Population: Full analysis set
Measure: Number; unit: Youden's index
Groups:
- All Participants: The analysis of whether progesterone level is a predictor for ongoing pregnancy used all participants.
Arm/Group | All Participants
Number analyzed (Participants) | 124
Youden's index
  Day 7 | 0.5189
  Day of hCG Administration (approx Day 10) | 0.4944

3. Secondary Outcome: Percentage of Participants With Ongoing Pregnancy
Description: Ongoing pregnancy is defined as having a positive foetal heart action nine or more weeks after the first positive pregnancy test.
Time Frame: approximately 3.5 months from study start (at least 9 weeks after first positive pregnancy test)
Population: The per-protocol (PP) set -- defined as participants of the full analysis set without any major protocol violation (i.e., any deviation which was likely to bias the assessment of the primary endpoint).
Measure: Number; unit: percentage of participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
percentage of participants | 29.2 | 31.0
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 1.00, Fisher Exact — The significance level is 0.05

4. Secondary Outcome: Number of Follicles at hCG Administration
Description: Number of follicles >=17 mm diameter detected by pelvic ultrasound examination at day of hCG administration.
Time Frame: approximately day 10
Population: The per-protocol (PP) set of participants with non-missing values. PP set is defined as participants of the full analysis set without any major protocol violation (i.e., any deviation which was likely to bias the assessment of the primary endpoint).
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 57
follicles | 8.7 (4.7) | 10.5 (4.1)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

5. Secondary Outcome: Average Follicle Diameter at hCG Administration
Time Frame: approximately day 10
Population: The per-protocol (PP) set of participants with non-missing values.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 57
mm | 17.6 (1.8) | 18.1 (1.2)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.121, t-test, 2 sided — The significance level is 0.05

6. Secondary Outcome: Number of Cumulus-oocyte Complexes Retrieved
Description: Cumulus-oocyte complexes are oocytes with surrounding cumulus cells.
Time Frame: approximately day 12 after study start
Population: The per-protocol (PP) set of participants with non-missing values.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 57
oocytes | 6.8 (4.2) | 10.0 (4.6)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Level of significance is 0.05

7. Secondary Outcome: Number of Pronuclear Oocytes
Description: Pronuclear oocytes are fertilized oocytes.
Time Frame: approximately day 13 after study start
Population: The per-protocol (PP) set of participants with non-missing values.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 57
oocytes | 3.7 (2.8) | 5.9 (3.7)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

8. Secondary Outcome: Number of Participants With Pronuclear Stage Oocytes at Each Quality Grade
Description: The count of participants with different quality grades of pronuclear stage oocytes is offered. Pronuclear stage oocytes are categorized into seven grades (0A, 0B, 1-5) representing different patterns of pronuclear morphology, according to the German Pronuclear Morphology Study Group. 0A is the highest quality oocyte and grade 5 is the lowest quality.
  Participants can have pronuclear stage oocytes of different grades and therefore are counted more than once.
Time Frame: approximately day 13
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
participants
  Grade 0A | 11 | 17
  Grade 0B | 15 | 23
  Grade 1 | 33 | 40
  Grade 2 | 15 | 25
  Grade 3 | 8 | 24
  Grade 4 | 2 | 11
  Grade 5 | 11 | 23

9. Secondary Outcome: Number of Embryos Transferred
Description: Mean number of embryos transferred 2-3 days following oocyte retrieval.
Time Frame: approximately day 14
Population: The per-protocol (PP) set who had embryos transferred. PP set is defined as participants of the full analysis set without any major protocol violation (i.e., any deviation which was likely to bias the assessment of the primary endpoint).
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 46 | 54
embryos | 2.0 (0.5) | 2.0 (0.4)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.482, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

10. Secondary Outcome: Best Quality of an Embryo Transferred
Description: Embryo quality was measured by the following grades:
  * Grade 1: Evenly sized cells, regular cleavage, no fragmentation
  * Grade 2: Regular or slightly irregular cleavage, <=20% fragmentation
  * Grade 2.5: Regular or slightly irregular cleavage, >20%and <=50% fragmentation
  * Grade 3: Irregular cleavage, >50% fragmentation, >1 intact cell
  * Grade 4: Extensive fragmentation, only 1 cell intact
  * Grade 5: Totally fragmented, no viable cells.
  Grade 1 represents the healthiest embryos and Grade 5 embryos are not viable.
Time Frame: approximately day 14
Population: Per protocol set of participants who had embryos transferred
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 46 | 54
participants
  Grade 1 | 22 | 26
  Grade 2 | 18 | 22
  Grade >2 | 6 | 6
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.871, Chi-squared — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

11. Secondary Outcome: Number of Frozen Oocytes at Pronuclear Stage
Description: No more than three normally developed embryos were transferred 2-3 days after oocyte retrieval. Other normally developed embryos were frozen.
Time Frame: approximately day 14
Population: Per protocol set of participants who had embryos transferred
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 46 | 54
oocytes | 1.0 (2.2) | 2.7 (2.9)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

12. Secondary Outcome: Endometrial Thickness on Day of hCG Administration
Description: Endometrial thickness was assessed by pelvic ultrasound on the day of hCG administration.
Time Frame: approximately day 10
Population: Per protocol set of participants. One participant in the Follitrophin Alpha arm was missing a measurement.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 57
mm | 10.8 (2.1) | 11.0 (2.2)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.620, t-test, 2 sided — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

13. Secondary Outcome: Estradiol (E2) Levels on Day of hCG Administration
Time Frame: approximately day 10
Population: Per protocol set. Five participants from each treatment arm were missing blood samples.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 43 | 53
ng/ml | 1.81 (1.21) | 1.65 (0.87)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.478, t-test, 2 sided — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

14. Secondary Outcome: Percentage of Participants With Successful Embryo Transfer
Time Frame: approximately day 18
Population: Per protocol set
Measure: Number; unit: percentage of participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
percentage of participants
  No | 4.2 | 6.9
  Yes | 95.8 | 93.1
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.69, Fisher Exact — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

15. Secondary Outcome: Number of Days Stimulated With Gonadotrophins
Description: Number of days in which gonadotrophins were administered until hCG criteria were met. If hCG criteria were not met by day 13, the participant was withdrawn from the study.
Time Frame: Day 1 up to Day 12
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
days | 8.7 (1.9) | 9.1 (1.6)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.295, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

16. Secondary Outcome: Number of Ampoules of Gonadotrophins Used
Description: Number of ampoules of gonadotrophins used with the goal of reaching hCG criteria. Each ampoule contained 75 IU of either menotrophin or follitrophin alpha.
Time Frame: Day 1 up to Day 12
Population: Per protocol set
Measure: Mean (Standard Deviation); unit: ampoules
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
ampoules | 20.8 (7.5) | 21.5 (6.8)
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 0.405, Wilcoxon (Mann-Whitney) — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

17. Secondary Outcome: Percentage of Participants With Clinical Pregnancy 6 Weeks After the First Positive Pregnancy Test
Description: A pelvic ultrasound scan was performed approximately 6 weeks after the first positive pregnancy test and the presence of an active foetal heart action indicated a clinical pregnancy.
Time Frame: approximately 2.5 months from start of study, 6 weeks after first positive pregnancy test
Population: Per protocol set
Measure: Number; unit: percentage of participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 48 | 58
percentage of participants | 29.2 | 31.0
Statistical Analysis 1: Comparison: Menotrophin vs Follitrophin Alpha; Test type: Superiority or Other; p = 1.000, Fisher Exact — The significance level is 0.05. P-values are not adjusted for multiple tests and have to be interpreted exploratively

18. Secondary Outcome: Summary of Pregnancy Outcome
Description: Pregnancy outcomes were reported at the optional long-term follow up visit.
Time Frame: up to 10 months
Population: Per protocol set of participants who reported information during the optional long-term follow up visit.
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitrophin Alpha
Number analyzed (Participants) | 14 | 16
participants
  Live birth | 13 | 16
  Ectopic pregnancy | 1 | 0
  Congenial abnormality | 0 | 1

ADVERSE EVENTS:
Time Frame: -Menotrophin: Day 1 up to Day 23. Treatment with investigational product (up to Day 12), plus residual drug effect-10.5 days -Follitropin: Day 1 up to Day 17. Treatment with comparator product (up to Day 12), plus residual drug effort-5 days.
Groups:
- Menotrophin: Menotrophin 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 13 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
- Follitrophin Alpha: Follitrophin alpha 150 IU (up to 300 IU) by subcutaneous injection once per day in the morning for up to 13 days until human chorionic gonadotropin (hCG) criteria are met. Pituitary down-regulation (cetrorelix), ovulation induction (choriongonadotropin), and luteal phase support (intravaginal progesterone) are administered the same way in both treatment arms.
Arm/Group | Menotrophin | Follitrophin Alpha
Serious Adverse Events (participants affected / at risk) | 2/62 | 0/62
Other Adverse Events (participants affected / at risk) | 43/62 | 45/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menotrophin (N=62) | Follitrophin Alpha (N=62)
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menotrophin (N=62) | Follitrophin Alpha (N=62)
Tachycardia (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 12
Nausea (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Injection site erythema (General disorders) | 10 | 7
Injection site pruritus (General disorders) | 9 | 7
Injection site pain (General disorders) | 7 | 5
Injection site reaction (General disorders) | 5 | 4
Injection site swelling (General disorders) | 4 | 5
Fatigue (General disorders) | 3 | 2
Injection site rash (General disorders) | 2 | 2
Injection site haemorrhage (General disorders) | 1 | 1
Injection site inflammation (General disorders) | 0 | 2
Chills (General disorders) | 1 | 0
Injection site warmth (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 11 | 13
Dizziness (Nervous system disorders) | 2 | 3
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 2
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 1
Breast discomfort (Reproductive system and breast disorders) | 1 | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Nipple pain (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Premature ovulation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor.

Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.